CLINICAL TRIAL: NCT06747338
Title: A Randomized, Controlled, Open-label, Multicenter, Phase III Clinical Trial to Compare the Efficacy and Safety of KN026 Combined With HB1801 ± Carboplatin Versus Trastuzumab Combined With Pertuzumab and Docetaxel ± Carboplatin in Neoadjuvant Treatment of Early or Locally Advanced HER2-positive Breast Cancer.
Brief Title: A Phase III Study of KN026 in Combination With HB1801 ± Carboplatin as Neoadjuvant Treatment for Early or Locally Advanced HER2-Positive Breast Cancer
Acronym: Neo-Healer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KN026-004
Record Dates: First submitted 2024-12-13; First posted 2024-12-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Early or Locally Advanced HER2-positive Breast Cancer
MeSH Terms: interventions — pertuzumab; Trastuzumab; Docetaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: In this randomized, controlled, open-label, multicenter phase 3 study, treatment-naive with HER2-positive breast cancer were randomly assigned (1:1) centrally and stratified by early (T2-3, N0-1, M0), locally advanced (T2-3, N2-3, M0; T4, any N, M0) breast cancer, hormone receptor status, and the planned use of Carboplatin. Participants received six cycles of:: KN026 combined with HB1801 ± Carboplatin (Experimental) or Trastuzumab plus Pertuzumab and Docetaxel ± Carboplatin (Active Comparator).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KN026 plus HB1801 ± Carboplatin (Experimental): KN026 HB1801 Carboplatin
  Interventions: Drug: KN026; Drug: HB1801
- Pertuzumab and trastuzumab plus docetaxel ± Carboplatin (Active Comparator): Pertuzumab Trastuzumab Docetaxel Carboplatin
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: Docetaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: KN026 — KN026
  Arms: KN026 plus HB1801 ± Carboplatin
Drug: HB1801 — HB1801
  Arms: KN026 plus HB1801 ± Carboplatin
Drug: Pertuzumab — Pertuzumab
  Arms: Pertuzumab and trastuzumab plus docetaxel ± Carboplatin
Drug: Trastuzumab — Trastuzumab
  Arms: Pertuzumab and trastuzumab plus docetaxel ± Carboplatin
Drug: Docetaxel — Docetaxel
  Arms: Pertuzumab and trastuzumab plus docetaxel ± Carboplatin
Drug: Carboplatin — Carboplatin
  Arms: Pertuzumab and trastuzumab plus docetaxel ± Carboplatin

SUMMARY:
This randomized, controlled, open-label, multicenter study will evaluate the safety and efficacy of KN026 in combination with HB1801 ± Carboplatin as neoadjuvant therapy in patients with early or locally advanced HER2-positive breast cancer.

DETAILED DESCRIPTION:
In this randomized, controlled, open-label, multicenter Phase III trial, treatment-naive patients with HER2-positive breast cancer were centrally randomized (1:1) and stratified by disease stage, hormone receptor status, and the planned use of Carboplatin. Participants received six cycles of: neoadjuvant therapy: KN026 combined with HB1801 ± Carboplatin (Experimental) or Trastuzumab plus Pertuzumab and Docetaxel ± Carboplatin (Active Comparator). The primary endpoint was pathological complete response (pCR) in the breast, evaluated in the intention-to-treat (ITT) population.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the experiment and sign the informed consent;
2. Aged >= 18 years;
3. Histologically and cytologically confirmed primary invasive carcinoma of the breast with early (T2-3, N0-1, M0) or locally advanced stage (T2-3, N2-3, M0; T4, any N, M0) (AJCC 8th Edition);
4. ECOG PS 0-1;
5. HER2 positive (HER2+++ by IHC or HER2++ by IHC and ISH+);
6. Agree to receive surgical treatment for breast cancer in the participating research unit when the surgical standard is reached after neoadjuvant therapy;
7. Adequate organ and bone marrow function (no blood transfusions or hematopoietic stimulating factor classes within 14 days prior to the test);
8. Women of childbearing potential and male participants with partners of childbearing potential must agree to use effective contraception (as defined by the protocol) by the participant and/or partner for the duration of the study treatment and for at least 3 months (Docetaxel and HB1801) or 7 months (Pertuzumab, trastuzumab, KN026, and Carboplatin) after the last dose of study drug;

Exclusion Criteria:

1. Inflammatory or bilateral breast cancer;
2. History of non-breast malignancies within the 3 years prior to study entry, except for carcinoma in situ of the cervix or breast, and basal cell and squamous cell carcinomas of the skin, etc.;
3. The researchers determine that there are contraindications for breast cancer surgery;
4. Participants who underwent primary lumpectomy and/or axillary lymph node dissection biopsy prior to randomization (except for diagnostic biopsy of primary breast cancer or surgery for benign breast tumors);
5. Any previous systemic chemotherapy, endocrine therapy or anti HER2 biological therapy or local radiotherapy for breast cancer;
6. Sensitivity to any of the study medications or any of the ingredients or excipients of these medications;
7. Participants with known allergies and/or contraindications to glucocorticoids;
8. Have a congenital or acquired immune deficiency (such as HIV infection); 9 . Serious cardiac or cardiovascular disease or condition; 10 Serious chronic or active infections requiring intravenous antimicrobial, antifungal, or antiviral therapy were present within 14 days prior to randomization.

11. Patients who had undergone major organ surgery (excluding biopsy) within 28 days before randomization and have not fully recovered.

12. Potent inhibitors or inducers of CYP3A4 were used within 14 days before randomization or continued use was required.

13. Being enrolled in other clinical trials (except for non-interventional clinical trials or a follow-up period in an interventional trial) or at randomization was less than 4 weeks from the end of the previous clinical trial (end of treatment).

14. Pregnant or lactating. 15. The existence of other conditions that may interfere with the participant's study procedures or that do not correspond to the participant's maximum benefit from participating in the study or to the findings of the imaging study, such as a history of neurological or mental illness, alcohol abuse, drug use or substance abuse, any other disease or condition of clinical significance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-12-16 (Estimated); Study Completion 2027-12-16 (Estimated)

PRIMARY OUTCOMES:
tpCR (BIRC, AJCC 8th) | Through study completion, an average of 1 year
  tpCR (ypT0/Tis ypN0) is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy.

SECONDARY OUTCOMES:
EFS (INV, RECIST v1.1) | Through study completion, an average of 1 year
  EFS event was defined as the time between the data of randomization and the date on which any of the following events: disease progression; breast cancer recurrence; death attributable to any cause.
tpCR (INV, AJCC 8th) | Through study completion, an average of 1 year
  Description: tpCR (ypT0/Tis ypN0) is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy.
bpCR (BIRC and INV, AJCC 8th) | Through study completion, an average of 1 year
  bpCR (ypT0/Tis) is defined as an absence of invasive neoplastic cells at microscopic examination of the tumor remnants after surgery following primary systemic therapy.
ORR (INV, RECIST v1.1) | After 2 cycles of chemotherapy (21 days as 1 cycle).
iDFS (INV, RECIST v1.1) | 3 years after surgery
  IDFS event was defined as the time between the date of non-invasive disease, such as the date of surgery, and the date of the first occurrence of any of the following events: breast cancer recurrence; death attributable to any cause
Frequency and severity of TEAE and SAE | After each cycle of chemotherapy (21 days as 1 cycle), up to 1 years.
Concentration of KN026 and HB1801 in serum | After each cycle of chemotherapy (21 days as 1 cycle), up to 6 cycles.
Incidence of KN026 Anti-drug antibody (ADA) and neutralizing antibody (Nab) (if applicable) | After each cycle of chemotherapy (21 days as 1 cycle), up to 6 cycles.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials Information Group, Shanghai, China